CLINICAL TRIAL: NCT03711786
Title: The Sub-Saharan Africa Regional Partnership (SHARP) for Mental Health Capacity Building
Brief Title: The Sub-Saharan Africa Regional Partnership for Mental Health Capacity Building
Acronym: SHARP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Ministry of Health, Malawi (Other Government); Kamuzu University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 18-2211; 1U19MH113202-01 (NIH)
Record Dates: First submitted 2018-01-12; First posted 2018-10-18 (Actual); Results first posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2022-08

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: 10 clinics will be randomized 1:1 to either a basic or enhanced implementation package to support integration of evidence-based depression treatment.
Masking Description: As randomization is at the clinic level and cannot be masked, participants, care providers, and investigators will not be masked to allocation.
  Outcome assessors do not need to know study arm, but it will be operationally difficult to blind them to whether a clinic is receiving the basic or enhanced implementation package.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Basic implementation package (Active Comparator): Ten Malawi non-communicable diseases clinics will be randomized 1:1 to one of two implementation strategies to be used for two years followed by a 12-month follow-up period.
  Interventions: Other: Basic implementation package
- Enhanced implementation package (Experimental): Ten Malawi non-communicable diseases clinics will be randomized 1:1 to one of two implementation strategies to be used for two years followed by a 12-month follow-up period.
  Interventions: Other: Enhanced implementation package

INTERVENTIONS:
Other: Basic implementation package — The basic implementation package will involve identifying an internal coordinator who is one of the full-time on-site providers at the clinic. The internal coordinator provides mentoring to peers and support to leadership in implementing the treatment program and aligning it with clinic priorities.
  Arms: Basic implementation package
Other: Enhanced implementation package — The enhanced implementation package will combine the internal coordinator with an external quality assurance committee. This committee will complete quarterly audits at the facility to evaluate compliance with the depression treatment protocol as well as providing high-level support in implementing the treatment program through clinical expertise and limited on-site presence.
  Arms: Enhanced implementation package

SUMMARY:
This is a 10-site cluster-randomized implementation science trial that compares two clinic-level implementation strategies to facilitate ongoing Ministry of Health efforts to scale up depression treatment within non-communicable diseases clinics in Malawi. Primary outcomes are clinical care indicators measured at the level of the visit (patient screened yes/no; depression treatment initiated if indicated yes/no; depression treatment algorithm followed at follow-up yes/no). Secondary outcomes are patient health outcomes measured at the level of the participant.

DETAILED DESCRIPTION:
This 10-site cluster-randomized implementation science trial compares the success of two clinic-level strategies in achieving high-quality integration of depression treatment into 10 non-communicable diseases (NCD) clinics in Malawi. Clinics are randomized 1:1 to one of two clinic-level implementation strategies: a basic strategy involving an internal coordinator, and an enhanced strategy combining the internal coordinator with an external quality assurance monitoring and supervision team. During a pre-randomization run-in period (months 1-5), all clinics receive the basic strategy. During a post-randomization intervention period (months 6-38), half of the clinics continue to receive the basic strategy and half receive the enhanced strategy. Visit-level data (for primary outcomes) and participant enrollment and follow-up (for secondary outcomes) are collected from all 10 clinics during the run-in and intervention periods.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet the following eligibility criteria will be invited to participate:

* Ages 18-65 years (antidepressant treatment considerations differ for those <18 or >65 years, and these age groups are expected to be very rare in the target clinics),
* Current or new patient receiving care for either hypertension or diabetes from a participating NCD clinic
* Elevated depressive symptoms (PHQ-9 score ≥5)

Exclusion Criteria:

Patients will be excluded if they have

* a history of bipolar or psychotic disorder, or show emergent threat of self-harm.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 946 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian W Pence, PhD, Principal Investigator — UNC-Chapel Hill
Locations (12):
- Malawi (12):
  - Chilumba Rural Hospital, Chilumba, Karonga
  - Karonga District Hospital, Karonga
  - MEIRU, Karonga
  - Kasungu District Hospital, Kasungu
  - Bwaila Hospital, Lilongwe
  - UNC Project Malawi, Lilongwe
  - Machinga District Hospital, Machinga
  - Mchinji District Hospital, Mchinji
  - Mulanje District Hospital, Mulanje
  - Phalombe Rural Health Center, Phalombe
  - Salima District Hospital, Salima
  - Zomba Central Hospital, Zomba

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared via the National Institute of Mental Health Data Archive. This will include de-identified individual-level data. Other researchers can apply to the National Institute of Mental Health Data Archive to access these data.
Time Frame: Data will be uploaded every 6 months. The first expected upload is on July 15, 2019.
Access Criteria: Access to the National Institute of Mental Health Data Archive is governed by the National Institute of Mental Health.
URL: https://nda.nih.gov/

REFERENCES:
- [Derived] Zimba CC, Malava JK, Mbota M, Matewere M, Akello H, Akiba CF, Landrum KR, Morrison A, Go V, Hosseinipour MC, Gaynes BN, Udedi M, Masiye J, Pence BW. Barriers and potential solutions for effective integration of depression care into non-communicable diseases clinics in Malawi: a qualitative end-point evaluation of the SHARP randomized controlled trial. Int J Ment Health Syst. 2025 Mar 6;19(1):8. doi: 10.1186/s13033-025-00663-z. PMID 40050899
- [Derived] Pence BW, Gaynes BN, Udedi M, Kulisewa K, Zimba CC, Akiba CF, Dussault JM, Akello H, Malava JK, Crampin A, Zhang Y, Preisser JS, DeLong SM, Hosseinipour MC. Two implementation strategies to support the integration of depression screening and treatment into hypertension and diabetes care in Malawi (SHARP): parallel, cluster-randomised, controlled, implementation trial. Lancet Glob Health. 2024 Apr;12(4):e652-e661. doi: 10.1016/S2214-109X(23)00592-2. Epub 2024 Feb 23. PMID 38408462
- [Derived] Sansbury GM, Pence BW, Zimba C, Yanguela J, Landrum K, Matewere M, Mbota M, Malava JK, Tikhiwa H, Morrison AM, Akiba CF, Gaynes BN, Udedi M, Hosseinipour MC, Stockton MA. Improving integrated depression and non-communicable disease care in Malawi through engaged leadership and supportive implementation climate. BMC Health Serv Res. 2023 Dec 14;23(1):1413. doi: 10.1186/s12913-023-10344-7. PMID 38098079
- [Derived] Zimba CC, Akiba CF, Matewere M, Thom A, Udedi M, Masiye JK, Kulisewa K, Go VF, Hosseinipour MC, Gaynes BN, Pence BW. Facilitators, barriers and potential solutions to the integration of depression and non-communicable diseases (NCDs) care in Malawi: a qualitative study with service providers. Int J Ment Health Syst. 2021 Jun 11;15(1):59. doi: 10.1186/s13033-021-00480-0. PMID 34116699
- [Derived] Gaynes BN, Akiba CF, Hosseinipour MC, Kulisewa K, Amberbir A, Udedi M, Zimba CC, Masiye JK, Crampin M, Amarreh I, Pence BW. The Sub-Saharan Africa Regional Partnership (SHARP) for Mental Health Capacity-Building Scale-Up Trial: Study Design and Protocol. Psychiatr Serv. 2021 Jul 1;72(7):812-821. doi: 10.1176/appi.ps.202000003. Epub 2020 Dec 9. PMID 33291973
- [Derived] Akiba CF, Zimba CC, Thom A, Matewere M, Go V, Pence B, Gaynes BN, Masiye J. The role of patient-provider communication: a qualitative study of patient attitudes regarding co-occurring depression and chronic diseases in Malawi. BMC Psychiatry. 2020 May 19;20(1):243. doi: 10.1186/s12888-020-02657-2. PMID 32429877

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ten clinics began the pre-randomization run-in period. All ten continued into the randomized intervention period. Primary outcomes (clinical care indicators) are measured at the level of the visit; visits do not overlap between the run-in and intervention periods. Secondary outcomes are measured at the level of the enrolled participant over 12 months of follow-up; enrolled participants do not overlap between the run-in and intervention periods. The numbers below represent participants.
Pre-assignment Details: 357 participants were enrolled during the run-in period before randomization. These participants are reported according to the arm to which their clinic was later assigned. 589 participants were enrolled during the intervention period post-randomization.
  By protocol, participants completed the study at 12 months post-consent. However, for logistical reasons the decision was made to conclude the study early and so the final 91 participants completed the study at 6 months.
Units Other Than Participants: Clinics
Groups:
- Basic Implementation Package: The basic implementation package is a clinic-level strategy that involves identifying an internal coordinator who is one of the full-time on-site providers at the clinic. The internal coordinator provides mentoring to peers and support to leadership in implementing the treatment program and aligning it with clinic priorities.
- Enhanced Implementation Package: The enhanced implementation package is a clinic-level strategy that combines the internal coordinator (basic arm) with an external quality assurance committee. This committee will complete quarterly audits at the facility to evaluate compliance with the depression treatment protocol as well as providing high-level support in implementing the treatment program through clinical expertise and limited on-site presence.
Period: Period 1: Recruited in Study Months 1-5
Arm/Group | Basic Implementation Package | Enhanced Implementation Package
Started | 168; 5 Clinics | 189; 5 Clinics
3-month Assessment | 162; 5 Clinics | 186; 5 Clinics
6-month Assessment | 156; 5 Clinics | 179; 5 Clinics
12-month Assessment | 148; 5 Clinics | 183; 5 Clinics
Completed | 148; 5 Clinics | 183; 5 Clinics
Not Completed | 20; 0 Clinics | 6; 0 Clinics
Not completed — Lost to Follow-up | 13 | 4
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Death | 7 | 1
Period: Period 1: Recruited in Study Months 6-32
Arm/Group | Basic Implementation Package | Enhanced Implementation Package
Started | 301; 5 Clinics | 288; 5 Clinics
3-month Assessment | 275; 5 Clinics | 264; 5 Clinics
6-month Assessment | 277; 5 Clinics | 267; 5 Clinics
12-month Assessment | 237; 5 Clinics | 220; 5 Clinics
Completed | 279; 5 Clinics | 258; 5 Clinics
Not Completed | 22; 0 Clinics | 30; 0 Clinics
Not completed — Lost to Follow-up | 17 | 21
Not completed — Withdrawal by Subject | 0 | 5
Not completed — Death | 5 | 4

BASELINE CHARACTERISTICS:
Population: Primary outcomes 1-3 are measured at the level of the medical visit (n=60,774 above). Secondary patient-reported outcomes 4-5 are measured at the level of the patient (n=946 above).
Units Other Than Participants: Medical Visits
Groups:
- Total: Total of all reporting groups
Arm/Group | Basic Implementation Package | Enhanced Implementation Package | Total
Number analyzed (Participants) | 469 | 477 | 946
Number analyzed (Medical Visits) | 27187 | 33587 | 60774
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 0 | 3
  Between 18 and 65 years | 456 | 462 | 918
  >=65 years | 10 | 15 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (9.9) | 50.5 (9.8) | 50.8 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 366 | 392 | 758
  Male | 103 | 85 | 188
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black African non-Hispanic | 469 | 477 | 946
Region of Enrollment [Count of Participants; unit: Participants]
  Malawi | 469 | 477 | 946

OUTCOME MEASURES:

1. Primary Outcome: Fidelity in Depression Screening: Number of Screening-eligible Visits at Which Depression Screening is Completed
Description: This primary outcome is measured at the level of the clinician-patient visit out of all clinic visits during the intervention period, including visits with both consented and non-consented patients. The outcome is based on aggregate clinic process data including number of visits for which the patient is not already engaged in depression treatment (denominator) and number of visits for which the patient is screened for depression (numerator) on each clinic day at each facility. Completion of depression screening (successful outcome) is defined as the clinician completing the Patient Health Questionnaire-2 (PHQ-2), and, if the PHQ-2 score is >0, also completing the PHQ-9 with the patient.
Time Frame: Measured based on data from clinic visits on each clinic day throughout study period
Population: The population for this outcome is all screening-eligible clinician-patient visits during the study period, not patient participants. Aggregate data are captured for visits with both consented and non-consented patients. The enrolled participants (n=301 and 288) constitute a small portion of all captured visits (n=27,187 and 33,587), but non-consented patients (who are not uniquely identified) represent a large portion.
Measure: Count of Units; unit: Visits
Units Other Than Participants: Visits
Arm/Group | Basic Implementation Package | Enhanced Implementation Package
Number analyzed (Participants) | 301 | 288
Number analyzed (Visits) | 27187 | 33587
Visits | 14712 | 15888
Statistical Analysis 1: Comparison: Basic Implementation Package vs Enhanced Implementation Package; Test type: Superiority; p = 0.836, Regression - GEE, logistic; From Wald z-statistic from generalized estimating equations (GEE) model with bias-corrected standard error; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.22 to 6.65] — Enhanced arm (index) compared to basic arm (referent). GEE model with bias-corrected standard errors

2. Primary Outcome: Fidelity in Depression Treatment Initiation: Number of Treatment-eligible Visits for Which Depression Treatment Actually Starts Within 30 Days of Identification
Description: This primary outcome is measured at the level of the clinician-patient visit out of all treatment-eligible visits during the intervention period, including visits with both consented and non-consented patients. The outcome is based on aggregate clinic process data including number of visits for which the patient is eligible for depression treatment (denominator) and number of visits for which the patient initiates depression treatment (numerator) on each clinic day at each facility. Eligible for depression treatment is defined as PHQ-9 total score of 5 or above. Initiating depression treatment is defined as prescription of antidepressant medication or referral to Friendship Bench psychosocial counselors within 30 days of positive screen.
Time Frame: Measured based on data from clinic visits on each clinic day throughout study period
Population: The population for this outcome is all depression treatment-eligible clinician-patient visits during the study period, not patient participants. Aggregate data are captured for visits with both consented and non-consented patients. The enrolled participants (n=301 and 288) constitute a portion of all captured visits for this outcome (n=610 and 545), but non-consented patients (who are not uniquely identified) represent an additional portion.
Measure: Count of Units; unit: Visits
Units Other Than Participants: Visits
Arm/Group | Basic Implementation Package | Enhanced Implementation Package
Number analyzed (Participants) | 301 | 288
Number analyzed (Visits) | 610 | 545
Visits | 601 | 538
Statistical Analysis 1: Comparison: Basic Implementation Package vs Enhanced Implementation Package; Test type: Superiority; p = 0.877, Regression - GEE, logistic; From Wald z-statistic from GEE model with bias-corrected standard error; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.12 to 6.14] — Enhanced arm (index) compared to basic arm (referent). GEE model with bias-corrected standard errors

3. Primary Outcome: Fidelity in Following the Depression Treatment Algorithm: Number of Treatment Follow-up Appointments in the First Three Months of Depression Treatment for Which the Clinical Treatment Decision Follows the Depression Treatment Guidelines
Description: This primary outcome is measured at the level of the clinician-patient visit out of all eligible visits during the intervention period. Eligible visits are clinical visits by consented participants within the first 90 days after initiating depression treatment. The outcome is based on clinic process data including number of clinic visits for which the participant is already engaged in depression treatment (denominator) and number of visits where the treatment decision follows the treatment algorithm (numerator) on each clinic day at each facility. Following the algorithm (positive outcome) is defined as: (1) if the participant has completed 6 counseling sessions, any action is acceptable; (2) otherwise, if the participant started counseling, either continuing counseling or starting medication; (3) if the participant started medication and PHQ-9 score <10, continuing medication; (4) if the participant started medication and PHQ-9 score >=10, continuing medication and increasing dose.
Time Frame: Within the first three months of follow-up after initiating depression treatment
Population: Population: all clinic visits for consented participants in the first 3 months after starting depression treatment. Analysis is restricted to consented participants because the clinic visit must be linked to information from the initial visit to define whether the treatment decision follows the algorithm. Participants may have multiple clinic visits during the three months. These are routine clinic visits and are not the 3-month research assessment referenced in the participant flow.
Measure: Count of Units; unit: Visits
Units Other Than Participants: Visits
Arm/Group | Basic Implementation Package | Enhanced Implementation Package
Number analyzed (Participants) | 74 | 69
Number analyzed (Visits) | 85 | 81
Visits | 14 | 69
Statistical Analysis 1: Comparison: Basic Implementation Package vs Enhanced Implementation Package; Test type: Superiority; p = 0.001, Regression - GEE, logistic; From Wald z-statistic from GEE model with bias-corrected standard error; Odds Ratio (OR) = 18.36, 95% CI 2-sided [3.23 to 104.23] — Enhanced arm (index) compared to basic arm (referent). GEE model with bias-corrected standard errors

4. Secondary Outcome: Number of Participants Achieving Depression Remission at 3 Months
Description: This secondary outcome is measured at the level of the consented participant. Depressive severity is determined using the Patient Health Questionnaire-9 (PHQ-9; range 0-27). The PHQ-9 is a self-reported questionnaire measuring depressive symptoms.This is a nine item measure with a response score for each item on a 4-point scale ranging from 0 (not at all) to 3 (nearly every day). Thus, the total score ranges from 0 to 27, with 0-4 indicating no depressive symptoms, 5-9 mild depression, 10-14 moderate depression, 15-19 moderately severe depression, and 20-27 severe depression. Depression remission is defined as a score <5.
Time Frame: Three months post enrollment
Population: All participants who completed the 3-month assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Basic Implementation Package | Enhanced Implementation Package
Number analyzed (Participants) | 275 | 264
Participants | 98 | 138
Statistical Analysis 1: Comparison: Basic Implementation Package vs Enhanced Implementation Package; Test type: Superiority; p = 0.017, Regression - GEE, logistic; From Wald z-statistic from GEE model with bias-corrected standard error; Odds Ratio (OR) = 2.15, 95% CI 2-sided [1.15 to 4.01] — Enhanced arm (index) compared to basic arm (referent). GEE model with bias-corrected standard errors

5. Secondary Outcome: Number of Participants With Well Controlled NCD at 3 Months
Description: This secondary outcome is measured at the level of the consented participant. Hypertension is measured by research assistants at each study visit while fasting blood glucose is measured as part of routine clinical care and will be abstracted. Well-controlled non-communicable disease (NCD) will be defined for hypertension patients as systolic blood pressure (BP) <140 mmHg AND diastolic blood pressure <90 mmHg, and for diabetes patients as fasting blood glucose <130 mg/dl, following the Malawi Clinical Guidelines for the Management of NCDs.
Time Frame: Three months post enrollment
Population: Analysis population restricted to those (1) completing 3-month assessment (n=275;264); (2) hypertension diagnosis at baseline (n=221;234); (3) completing 3-month in person (n=59;90). Item 2 above is to exclude participants who only had a diabetes diagnosis at baseline because blood glucose measures were not consistently available from clinical records. Item 3 above is because with COVID, most follow-ups moved to phone in which case BP was no longer collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Basic Implementation Package | Enhanced Implementation Package
Number analyzed (Participants) | 59 | 90
Participants | 35 | 51
Statistical Analysis 1: Comparison: Basic Implementation Package vs Enhanced Implementation Package; Test type: Superiority; p = 0.759, Regression - GEE, logistic; From Wald z-statistic from GEE model with bias-corrected standard error; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.45 to 1.80] — Enhanced arm (index) compared to basic arm (referent). GEE model with bias-corrected standard errors

ADVERSE EVENTS:
Time Frame: Adverse events were collected from consent through each participant's study completion, up to approximately 12 months post-consent.
Description: Deaths were assessed systematically for any participant lost to contact through consultation of clinical records and community tracing. Hospitalizations and suicidal ideation were queried systematically at each research assessment.
Arm/Group | Basic Implementation Package | Enhanced Implementation Package
All-Cause Mortality (participants affected / at risk) | 12/469 | 5/477
Serious Adverse Events (participants affected / at risk) | 31/469 | 11/477
Other Adverse Events (participants affected / at risk) | 54/469 | 90/477
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Basic Implementation Package (N=469) | Enhanced Implementation Package (N=477)
Abdominal pain - Hospitalization (Gastrointestinal disorders) | 1 (2) | 0 (0)
Anaemia - Hospitalization (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Asthma - Hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Broken leg - Hospitalization (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Constipation - Hospitalization (Gastrointestinal disorders) | 1 (1) | 0 (0)
Convulsions - Hospitalization (Nervous system disorders) | 0 (0) | 1 (1)
Diarrhea - Hospitalization (Gastrointestinal disorders) | 0 (0) | 1 (1)
Elevated blood pressure - Hospitalization (Metabolism and nutrition disorders) | 10 (11) | 4 (4)
Emphysema - Hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epilepsy - Hospitalization (Nervous system disorders) | 1 (1) | 0 (0)
Hyperglycemia - Hospitalization (Endocrine disorders) | 11 (13) | 4 (4)
Hypoglycemia - Hospitalization (Endocrine disorders) | 5 (5) | 0 (0)
Jaundice - Hospitalization (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Low blood pressure - Hospitalization (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malaria - Hospitalization (Infections and infestations) | 3 (3) | 1 (1)
Physical therapy referral - Hospitalization (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatism - Hospitalization (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Basic Implementation Package (N=469) | Enhanced Implementation Package (N=477)
Suicidal ideation (Psychiatric disorders) | 54 (57) | 90 (106) — Any thoughts of self-harm or being better off dead in the past two weeks, as assessed by question 9 of the Patient Health Questionnaire-9.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-11): https://cdn.clinicaltrials.gov/large-docs/86/NCT03711786/Prot_SAP_000.pdf